CLINICAL TRIAL: NCT03787030
Title: Application of Vitamin E Acetate Ointment vs Nitroglycerin Ointment for the Treatment of Chronic Anal Fissure
Brief Title: Application of Vitamin E on Anal Fissure
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hospital General Universitario Elche (Other)
Responsible Party: Principal Investigator, Jaime Ruiz-Tovar, MD, PhD, Department of Surgery, Hospital General Universitario Elche
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Garcia 2018-12
Record Dates: First submitted 2018-12-21; First posted 2018-12-26 (Actual); Last update posted 2020-04-22 (Actual); Status verified 2020-04

CONDITIONS: Pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: A nurse blinded to the treatment applied will evaluate the healing of chronic anal fissure and quantify pain
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vitamin E acetate (Experimental): Commercially available plastic tubes containing vitamin E acetate ointment (Filme Olio, Hulka SRL, Italy) were purchased from pharmacies. The dosage for all the patients was 1ml of ointment (containing 1100% vitamin E), applied with a gloved finger to the distal anal canal, every 12 hours for an 8-week period.
  Interventions: Drug: Vitamin E Acetate ointment
- Glyceryl trinitrate ointment (Active Comparator): Commercially available aluminium tubes containing 0.4 glyceryl trinitrate ointment (Rectogesic, proStrakan Group, Galashiels, UK) were purchased from pharmacies. The dosage for all the patients was 375 mg of ointment (containing 1.5 mg of glyceryl trinitrate), applied with a gloved finger to the distal anal canal, every 12 hours for an 8-week period.
  Interventions: Drug: Glyceryl trinitrate ointment

INTERVENTIONS:
Drug: Vitamin E Acetate ointment — Application of 1 ml of ointment to the distal anal canal, every 12 hours for an 8-week period.
  Arms: Vitamin E acetate
Drug: Glyceryl trinitrate ointment — Application of 375 mg of ointment to the distal anal canal, every 12 hours for an 8-week period.
  Arms: Glyceryl trinitrate ointment

SUMMARY:
Patients were randomized into 2 groups:

* Vitamin E: Vitamin E ointment will be applied during 8 weeks
* Nitroglycerin: Nitroglycerin ointment will be applied during 8 weeks

Healing rate of chronic anal fissure in patients receiving Nitroglycerin ointment and subjects patients receiving Vitamin E ointment were evaluated .

DETAILED DESCRIPTION:
Patients were randomly assigned to experimental and control groups: those patients receiving vitamin E ointment (Experimental Group - EG) and those receiving glyceryl trinitrate ointment (Control Group - CG).

Treatments:

Glyceryl trinitrate ointment (GTO): Commercially available aluminium tubes containing 0.4 glyceryl trinitrate ointment (Rectogesic, proStrakan Group, Galashiels, UK) were purchased from pharmacies. The dosage for all the patients was 375 mg of ointment (containing 1.5 mg of glyceryl trinitrate), applied with a gloved finger to the distal anal canal, every 12 hours for an 8-week period.

Vitamin E acetate ointment (VEA): Commercially available plastic tubes containing VitaminE acetate ointment (Filme Olio, Hulka SRL, Italy) were purchased from pharmacies. The dosage for all the patients was 1ml, applied with a gloved finger to the distal anal canal, every 12 hours for an 8-week period.

Healing rate of chronic anal fissure was investigated.

ELIGIBILITY:
Inclusion Criteria:

* Patients with diagnosis of chronic anal fissure

Exclusion Criteria:

* patients with associated anal pathologies
* intestinal inflammation disorders
* immunosuppression
* fissures secondary to underlying diseases (eg, AIDS, tuberculosis, or sexually transmitted diseases)
* patients with a history of headaches, heart disease, or intolerance to nitrates
* pregnant or lactating women
* patients with closed angle glaucoma

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2018-12-21 (Actual); Primary Completion 2019-02-28 (Actual); Study Completion 2019-02-28 (Actual)

PRIMARY OUTCOMES:
Pain associated to anal fissure: Visual Analogic Scale | 8 weeks
  Pain will be evaluated after finishing the treatment, by a Visual Analogic Scale, ranging from 0 (absence of pain) to 100mm (unbearable pain)

SECONDARY OUTCOMES:
Number of participants achieving the healing of the fissure | 8 weeks
  Healing, defined as evidence of fissure reepithelization

CONTACTS AND LOCATIONS:
Overall Officials: Carolina Llavero, Study Director — Garcilaso Clinic
Locations (1):
- Garcilaso Clinic, Madrid, Spain

REFERENCES:
- [Derived] Ruiz-Tovar J, Llavero C. Perianal Application of Glyceryl Trinitrate Ointment Versus Tocopherol Acetate Ointment in the Treatment of Chronic Anal Fissure: A Randomized Clinical Trial. Dis Colon Rectum. 2022 Mar 1;65(3):406-412. doi: 10.1097/DCR.0000000000002120. PMID 34803148